CLINICAL TRIAL: NCT06397105
Title: Boosting Refugee Integration Through Psychological Intervention (BRIGHT) - a Pilot Randomised Controlled Trial
Brief Title: Feasibility and Acceptability of BRIGHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: ETH Zurich (Other); The University of New South Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BASEC-2023-00857-pilot
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Psychological Distress; PTSD; Trauma, Psychological
Keywords: Problem Management Plus; Psychological Distress; Mental Health Care; Refugees
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychological Trauma

STUDY DESIGN:
Intervention Model Description: The pilot RCT will inform us about the feasibility of PM+ under usual practice conditions.
Who Masked: Outcomes Assessor
Masking Description: All instruments and questions of the screening and baseline assessment will be assessed as an assisted self-assessment in the presence of a trained assessor fluent in the participant's mother tongue blind to the allocation status of the participants.The follow-up assessments are administered either as an online self-assessment, as an assisted online self-assessment or as an self-assessment in presence. In either case, the trained assessors are blind to the allocation status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Problem Management Plus (Experimental): The participants who are assigned to the intervention group will receive five sessions of PM+, a psychological intervention which has been developed by the WHO. PM+ is a short, transdiagnostic (i.e., not specifically aimed at treating a certain mental disorder) program aiming to reduce common mental health symptoms and improve psychosocial functioning. In addition, participants will receive three telephone booster sessions and will have access to a digital support program.
  Interventions: Behavioral: Problem Management Plus
- waitlist control group (Other): The control group will receive the augmented PM+ intervention 12 months after the baseline assessment.
  Interventions: Behavioral: Problem Management Plus
- observational control group (No Intervention): Participants who scored below 20 on the K10 will will only be part of the baseline assessments and receive no intervention.

INTERVENTIONS:
Behavioral: Problem Management Plus — Problem Management Plus (PM+) is a brief, psychological intervention program based on CBT techniques that are empirically supported and formally recommended by the WHO. The full protocol was developed by the WHO and the University of New South Wales, Australia. The manual involves the following empirically supported elements: problem solving plus stress management, behavioural activation, facing fears, and accessing social support. These elements have been recommended in recent WHO guidelines.
  Additionally, the original five PM+ sessions will be augmented in two ways. First, the participants will receive three 30-45-minutes telephone booster sessions 10, 22, and 34 weeks after the final original PM+ session. The second augmentation strategy will comprise a digital support program that participants can access via the internet.
  Arms: Problem Management Plus; waitlist control group

SUMMARY:
Refugees and asylum seekers (RAS) face numerous stressors and adversities which put them at risk for developing mental health problems. However, access to adequate mental health care in host countries is limited. To address this problem, the World Health Organization (WHO) introduced Problem Management Plus (PM+), a short, low-intensity psychological intervention administered by non-professionals, aiming to alleviate common mental disorders among crisis-affected communities.

The objective of this pilot RCT is to assess the feasibility and acceptability of an adapted version of PM+ for refugees and asylum-seekers. This will inform the design of a definitive RCT and implementation study.

DETAILED DESCRIPTION:
Refugees and asylum seekers (RAS) are often exposed not only to potentially traumatic events before and during migration but also to significant post-migration stressors. Due to this combined burden, RAS are at increased risk for developing mental health problems. In accessing mental health care in the host countries, however, they face several barriers including waitlists, stigma and communication difficulties. Consequently, RAS are frequently underdiagnosed and often do not receive adequate medical treatment despite an urgent need.

To improve the access to evidence-based psychological interventions, the WHO developed a series of scalable interventions. One of these is Problem Management Plus (PM+), a brief, low-intensity psychological intervention, delivered by paraprofessionals, that addresses common mental disorders in people affected by adversity. PM+ consists of 5 sessions that comprise evidence-based techniques of (a) problem solving, (b) stress management, (c) behavioral activation, and (d) accessing social support. The present study aims at expanding the existing PM+ intervention by providing additional booster sessions and access to a digital support program.

PM+ has been proven to be an effective method for reducing mental health problems and improving the psychosocial functioning of people in crisis in various countries and contexts, including Switzerland.

Despite its effectiveness, far too little attention has been paid to the successful implementation of such low-intensity psychological interventions into real-world health care systems.

The present pilot RCT aims to investigate the feasibility and acceptability of an augmented version of PM+ for refugees and asylum-seekers to inform a full-scale, definitive randomized controlled trial and implementation study. Data will be collected regarding the feasibility and acceptability of all study components, including recruitment, drop-out rate, protocol adherence, study visit attendance and the time burden of parent questionnaires. These data will inform the design of a full scale randomized controlled trial to evaluate the efficacy of augmented PM+ in refugees and asylum-seekers.

ELIGIBILITY:
Inclusion Criteria:

* refugees and asylum seekers (RAS) aged 16 or older;
* residing in one of the participating local sites (Swiss municipalities, namely, Gemeinden, and transitional asylum centers, namely, Durchgangszentren) where PM+ is offered and which gave their consent for participation in the RCT;
* speaking at least one of the following 12 languages: German, English, French, Arabic, Farsi, Kurdish, Tigrinya, Turkish, Ukrainian, Russian, Tamil, and Pashto;
* obtaining a score of 20 or higher on the Kessler Psychological Distress Scale (K10; Kessler et al., 2002), a brief clinically validated screening questionnaire that assesses general psychological distress in the past 30 days. A score equal to or higher than 20 is used as an indication of moderate to high levels of psychological distress.

Exclusion Criteria:

* significant cognitive or neurological impairment measured through specific tools developed by the WHO and integrated into the PM+ manual (impairment questionnaire);
* acute medical conditions or severe mental disorders (e.g., psychotic or substance-abuse disorders) measured through specific tools developed by the WHO and integrated into the PM+ manual (impairment questionnaire);
* acute risk of suicide as measured by the Suicidal Ideation Attribution Scale (SIDAS; van Spijker et al., 2014) and the Thoughts of Suicide Questionnaire (World Health Organization WHO, 2016).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in psychological distress | Baseline assessment, 3 month FU assessment (3 months after baseline)
  Change in psychological distress will be measured with the Hopkins Symptom Checklist (HSCL-25). Items are rated on a scale from 1 to 4. Higher scores indicate more pronounced symptom severity.

SECONDARY OUTCOMES:
Change in posttraumatic stress disorder symptoms | Baseline assessment, 3 month FU assessment (3 months after baseline), 6 month FU assessment (6 months after baseline), 12 months FU assessment
  Change in posttraumatic stress disorder symptoms will be assessed using the 4-item short form of the PCL-5. Items are rated on a scale from 0 to 4 with higher scores indicating more pronounced symptom severity.
General psychological distress | Screening, 3 month FU assessment (3 months after baseline), 6 month FU assessment (6 months after baseline), 12 months FU assessment
  General psychological distress will be measured with the Kessler Psychological Distress Scale - K10 (Kessler et al., 2002), a brief screening questionnaire assessing general psychological distress in the past 30 days. It consists of ten items (e.g., "During the last 30 days, about how often did you feel tired out for no good reason?") rated on a 5-point Likert scale (1 = "none of the time" to 5 = "all of the time"), before summation (range 10-50).
Somatic symptoms | Baseline assessment, 3 month FU assessment (3 months after baseline), 6 month FU assessment (6 months after baseline), 12 months FU assessment
  Somatic symptoms will be assessed using the Somatic Symptom Scale (SSS-8). Items are rated on a scale from 0 to 4 with higher scores indicating higher symptom severity.
Reduction of post-migration stressors | Baseline assessment, 3 month FU assessment (3 months after baseline), 6 month FU assessment (6 months after baseline), 12 months FU assessment
  Changes in post-migration stressors will be assessed using a 9-item version of the Post Migration Living Difficulties Checklist (PMLDC). Items are rated on a scale from 0 to 4 with lower scores representing fewer post-migration stressors.
Exposure to potentially traumatic events | Baseline assessment
  Exposure to potentially traumatic events is indexed using a list of seven traumatic experiences. Overall trauma exposure is represented by a count of the number of traumatic event types (ranging from 0 to 7) experienced by each participant; higher scores indicate experience of more forms of traumatic events.
Level of integration | Baseline assessment, 6 month FU assessment (6 months after baseline), 12 months FU assessment
  Level of integration will be measured using the Immigration Policy Lab Integration Index (IPL-24). Items are rated between one and five points. Higher scores indicate more pronounced symptom severity.
Suicidal Ideation | Baseline assessment, 6 month FU assessment (6 months after baseline), 12 months FU assessment
  Suicidal Ideation is measured using the Suicidal Ideation Attribution Scale (SIDAS), a brief measure of severity of suicidal ideation assessing frequency, controllability, closeness to attempt, level of distress associated with the thoughts and impact on daily functioning. It consists of five items rated on a 11-point scale (0 = "Never" to 10 = "Always").
Change in psychological distress | 6 month FU assessment (6 months after baseline), 12 months FU assessment
  Change in psychological distress will be measured with the Hopkins Symptom Checklist (HSCL-25). Items are rated on a scale from 1 to 4. Higher scores indicate more pronounced symptom severity.
Feasibility of PM+ by the number of dropouts | Baseline assessment, 3 month FU assessment (3 months after baseline), 6 month FU assessment (6 months after baseline), 12 months FU assessment
  Monitoring of the dropouts by number of participants

CONTACTS AND LOCATIONS:
Overall Officials: Naser Morina, PD Dr., Principal Investigator — Klinik für Konsiliarpsychiatrie und Psychosomatik
Locations (1):
- Klinik für Konsiliarpsychiatrie und Psychosomatik, Universitätsspital Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spaaij J, Kiselev N, Berger C, Bryant RA, Cuijpers P, de Graaff AM, Fuhr DC, Hemmo M, McDaid D, Moergeli H, Park AL, Pfaltz MC, Schick M, Schnyder U, Wenger A, Sijbrandij M, Morina N. Feasibility and acceptability of Problem Management Plus (PM+) among Syrian refugees and asylum seekers in Switzerland: a mixed-method pilot randomized controlled trial. Eur J Psychotraumatol. 2022 Jan 31;13(1):2002027. doi: 10.1080/20008198.2021.2002027. eCollection 2022. PMID 35126880
- [Background] de Graaff AM, Cuijpers P, Twisk JWR, Kieft B, Hunaidy S, Elsawy M, Gorgis N, Bouman TK, Lommen MJJ, Acarturk C, Bryant R, Burchert S, Dawson KS, Fuhr DC, Hansen P, Jordans M, Knaevelsrud C, McDaid D, Morina N, Moergeli H, Park AL, Roberts B, Ventevogel P, Wiedemann N, Woodward A, Sijbrandij M; STRENGTHS Consortium; STRENGTHS consortium. Peer-provided psychological intervention for Syrian refugees: results of a randomised controlled trial on the effectiveness of Problem Management Plus. BMJ Ment Health. 2023 Feb;26(1):e300637. doi: 10.1136/bmjment-2022-300637. Epub 2023 Feb 8. PMID 36789918
- [Background] Dawson KS, Bryant RA, Harper M, Kuowei Tay A, Rahman A, Schafer A, van Ommeren M. Problem Management Plus (PM+): a WHO transdiagnostic psychological intervention for common mental health problems. World Psychiatry. 2015 Oct;14(3):354-7. doi: 10.1002/wps.20255. No abstract available. PMID 26407793
- [Background] Steel Z, Chey T, Silove D, Marnane C, Bryant RA, van Ommeren M. Association of torture and other potentially traumatic events with mental health outcomes among populations exposed to mass conflict and displacement: a systematic review and meta-analysis. JAMA. 2009 Aug 5;302(5):537-49. doi: 10.1001/jama.2009.1132. PMID 19654388